CLINICAL TRIAL: NCT05306561
Title: A Single Arm, Single Center Phase 4 Study to Evaluate Impact of a Single Systane iLux MGD Treatment Device Thermal Pulsation Treatment on Contact Lens Wearing Time and Tolerability, Meibomian Gland Secretion Scores, and Subjective Dry Eye Symptoms in Soft Contact Lens Wearing Subjects With Meibomian Gland Dysfunction
Brief Title: Evaluating Impact of Systane iLux on Dryness Symptoms and Wearing Time in Contact Lens Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Periman Eye Institute (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEI-IIT-70111343
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
Keywords: dry eye disease; meibomian gland dysfunction; ilux; thermal pulsation; contact lens
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Single arm trial
  Interventions: Procedure: Systane iLux thermal pulsation treatment

INTERVENTIONS:
Procedure: Systane iLux thermal pulsation treatment — Systane iLux thermal pulsation uses light emitting diode (LED) technology to emit light that is absorbed by pigments (melanin and hemoglobin) in the eyelid. The pigments convert the light energy to heat, which is then transferred to the surrounding tissues, including the meibomian glands. The device heats the eyelid to 40-42°C and maintains it above 40°C during the heating period, which can be 40 seconds or more. This helps melt the meibum. After the heating phase, the meibomian glands are expressed with the built in expression system.

SUMMARY:
To evaluate dry eye symptoms and contact lens wearing times after a single iLux treatment by evaluating change from baseline in OSDI scores, subjective CLDEQ8 and CL wearing time questionnaires, and meibomian gland secretion scores.

DETAILED DESCRIPTION:
A single arm, single center phase 4 study to evaluate impact of a single Systane iLux MGD Treatment Device thermal pulsation treatment on contact lens wearing time and tolerability, meibomian gland secretion scores, and subjective dry eye symptoms in soft contact lens wearing subjects with meibomian gland dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible subjects must be 18 years of age or older
2. Eligible subjects must be willing and able to provide an English language written Informed Consent Form
3. Be a current soft contact lens wearer for at least 2-18 hours a day 4-7 days a week but experiencing contact lens discomfort that limits the number of hours of comfortable contact lens wear.
4. Have worn the same commercially available soft contact lens (material, base curve, diameter) for the previous 90 days
5. Have new contact lens to wear starting the first day after iLux treatment
6. Have an OSDI score greater than ≥ 12
7. Have a CLDEQ8 score ≥ 12
8. Have a minimum meibomian gland expression score ≤ 12 (using MGD scoring system: apply pressure with korb expressor to 15 glands of lower lid (5 nasal, 5 central, 5 temporal): each gland will be scored from 0 to 3 (0 = no secretion, 1 = inspissated, 2 = cloudy, 3 = clear liquid), sum of score from each gland with equal total score, total score will range from 0-45.
9. Be able and willing to follow instructions and participate in all trial assessments and visits
10. Eligible subjects must be fully vaccinated against COVID-19

Exclusion Criteria:

1. Have any clinically significant slit-lamp findings at Visit 1 that in the opinion of the investigator may interfere with trial parameters
2. Have abnormal lid anatomy eg. entropion, ectropion or active lid lesion eg. hordeolum, chalazion that may interfere with administering iLux treatment
3. Had Lipiflow, iLux, Tear Care or manual meibomian gland expression in the last 30 days
4. Be a woman who is pregnant, nursing, or planning a pregnancy
5. Had ocular surgery within the last 90 days
6. Have used topical cyclosporine, lifitegrast, topical or facial steroids, serum tears, or oral doxycycline or tetracycline within the last 30 days before Visit 1
7. Had Intense Pulsed Light (IPL) treatment within last 30 days
8. Have active ocular infection or inflammation
9. Be a current wearer of extended wear contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with improvment in OSDI Questionnaire score from baseline to 1 month | 1 month
  OSDI (Ocular Surface Disease Index) is a subjective dry eye symptom questionnaire. A lower OSDI score represents less frequent and/or less severe symptoms.
Percentage of subjects with improvement in CLDEQ8 Questionnaire score from baseline to 1 month | 1 month
  CLDEQ8 (Contact Lens Dry Eye Questionnaire) is a subjective contact lens discomfort and dryness questionnaire. A lower CLDEQ8 score represents less frequent and/or less severe symptoms
Percentage of subjects with improvement in MGSS from baseline to 1 month | 1 month
  MGSS (Meibomian gland secretion score). To determine the meibomian gland score, secretion characteristics of 15 meibomian glands along the lower eyelid were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/ toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range between 0 and 45. A higher score reflects less meibomian gland dysfunction.
Percentage of subjects with improvement in comfortable SCL (soft contact lens) wearing time from baseline to 1 month | 1 month
  Total comfortable soft contact lens wearing time per week will be asked via questionnaire.
Percentage of subjects with dryness symptoms who reported wearing their contact lenses longer, 1 month post treatment. | 1 month
  Total soft contact lens wearing time per week will be asked via questionnaire.

SECONDARY OUTCOMES:
Mean change in Sodium Fluorescein and Lussamine Green staining from baseline to 1 month | 1 month
  Mean change in ocular surface staining (sodium fluorescein and lissamine green) from baseline as measured by the National Eye Institute and Oxford grading scales.
Mean change in TBUT from baseline to 1 month | 1 month
  The investigator instilled sodium fluorescein into the lower eyelid and asked the patient to blink several times, then stop. The time between the last blink and the first appearance of a dark spot on the cornea (formation of a dry area) on the otherwise continuously stained tear film was recorded in seconds. 3 consecutive measurements were taken, with TBUT defined as the average of the 3 measurements. A positive change value represents A positive change value represents a more stable tear film (improvement). Eyes were assessed individually.

CONTACTS AND LOCATIONS:
Locations (1):
- Periman Eye Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No